CLINICAL TRIAL: NCT05825430
Title: Direct Versus Ultrasound Guided PECS Block Effect on Controlling Postmastectomy Pain: A Prospective, Randomized, Single Blinded, Controlled Study.
Brief Title: Direct Versus US Guided PECS Block on Controlling Postmastectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC.5.1.2023
Record Dates: First submitted 2023-04-09; First posted 2023-04-24 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Postmastectomy Pain
Keywords: Ultrasound guided pecs block; Direct pecs

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): Patients will not receive any block
  Interventions: Drug: general anaesthetic technique only
- Direct pecs block group (Experimental): Pec I block will be given with 10 ml bupivacaine 0.25% which injected between two pectoral muscles and pecs II block will be given with 20 ml bupivacaine 0.25%.which given between pectoralis minor muscle and serratus muscle. Patients will receive direct pecs block by surgeon after closure of pectoralis muscle under direct vision and before skin closure.
  Interventions: Procedure: Direct pecs block
- Ultrasound guided pecs (Experimental): Pec I block will be given with 10 ml bupivacaine 0.25% which injected between two pectoral muscles and pecs II block will be given with 20 ml bupivacaine 0.25%.which given between pectoralis minor muscle and serratus muscle. Patients will receive ultrasound guided pecs block done after induction and before skin incision.
  Interventions: Procedure: Ultrasound guided pecs block

INTERVENTIONS:
Procedure: Direct pecs block — Patients will receive direct PECS block by surgeon after closure of pectoralis muscle under direct vision and before skin closure.
  All patients will receive the same general anaesthetic technique: In the form of iv induction by propofol 2mg /kg ,fentanyl 2 mic/ kg and intubation will be facilitated by atracurium 0.5 mg/kg. Anaesthesia will be maintained by isoflurane 1.5 MAC and incremental doses of atracurium 0.15 mg/kg every 20 min. At the end of surgery neuromuscular blocker reversed by neostigmine 50 micg/kg + atropine 20 micg /kg i.v.
  Other Names: 10 ml bupivacaine 0.25%
  Arms: Direct pecs block group
Procedure: Ultrasound guided pecs block — Patients will receive ultrasound guided pecs block after induction and before skin incision.
  All patients will receive the same general anaesthetic technique: In the form of iv induction by propofol 2mg /kg ,fentanyl 2 mic/ kg and intubation will be facilitated by atracurium 0.5 mg/kg. Anaesthesia will be maintained by isoflurane 1.5 MAC and incremental doses of atracurium 0.15 mg/kg every 20 min. At the end of surgery neuromuscular blocker reversed by neostigmine 50 micg/kg + atropine 20 micg /kg i.v.
  Other Names: 10 ml bupivacaine 0.25%
  Arms: Ultrasound guided pecs
Drug: general anaesthetic technique only — All patients will receive the same general anaesthetic technique: In the form of iv induction by propofol 2mg /kg ,fentanyl 2 mic/ kg and intubation will be facilitated by atracurium 0.5 mg/kg. Anaesthesia will be maintained by isoflurane 1.5 MAC and incremental doses of atracurium 0.15 mg/kg every 20 min. At the end of surgery neuromuscular blocker reversed by neostigmine 50 micg/kg + atropine 20 micg /kg i.v.
  Arms: Control group

SUMMARY:
Perioperative analgesia for surgery in carcinoma breast utilizes significant quantities of opioids as compared to cosmetic breast surgeries. Regional anesthesia reduces the need for perioperative opioids and thus may improve the outcome. The investigators decided to perform the modified pectoral nerve block ( Pec II) under vision after resection of tumor, without ultrasound and compare the postoperative analgesic and opioid sparing effects of the nerve block with ultrasound guided modified pectoral nerve block (Pec) in patients undergoing modified radical mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 50 years
* ASA I or II undergo elective simple mastectomy

Exclusion Criteria:

* patients with diabetes mellitus i
* Intradialytic hypotension,
* chronic kidney disease and Bronchial Asthma

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperative
  the amount of total postoperative morphine consumption

SECONDARY OUTCOMES:
postoperative visual analogue scale (VAS) | 24 hours postoperatively
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 "no pain" and 10 "worst pain.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Haney Baumey, Banhā
  - Neveen Kohaf, Tanta

IPD SHARING:
Plan to Share IPD: Yes
Data could be shared upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP, CSR